CLINICAL TRIAL: NCT01564511
Title: Effects of Electromechanical Gait Trainer on Endurance, Fatigue and Daily Life Autonomy in Patients With Multiple Sclerosis: a Randomized Control Trial
Brief Title: Effects of Electromechanical Gait Trainer in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, Prof. Smania Nicola, Universita di Verona
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: GT&SM-01
Record Dates: First submitted 2012-03-14; First posted 2012-03-27 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Robotic Rahabilitation; Fatigue; Gait disorder
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis; Fatigue; Mobility Limitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gait trainer treatment (Experimental): Roboti gait training by mean of Gangtrainer I
  Interventions: Device: Gait trainer treatment
- Conventional group (Sham Comparator): Convetional physical gait training
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Device: Gait trainer treatment — Patients will be subjected to 40 minutes of repetitive locomotor therapy on the Gait Trainer (GTI) (Reha-Stim, Berlin, Germany), followed by 10 minutes of passive joint mobilization and stretching exercises. The first 40 min session will be divided as follow: 15 min gait training; 5 minutes at rest; 15 minutes gait training; 5 minutes at rest. The GT-I consists of a double crank and rocker gear system, composed of two footplates positioned on two bars (coupler), two rockers, and two cranks that provide the propulsion.
  Arms: Gait trainer treatment
Other: Conventional treatment — The control group will be subjected to a conventional treatment that will consist of three different sets of exercises: 1) passive joint mobilization and stretching of lower limb muscles; 2) muscle strengthening exercises; 3) gait exercises. Each set of exercises lasted 10, 15 and 15 min, respectively with 2,5 min at rest between each set for a total of 40 minutes.
  Arms: Conventional group

SUMMARY:
Multiple Sclerosis is a very disabling disorder in young adult patients leading to an important limitation in daily life activities and social participation. Among of the different causes of disability in MS patients gait impairments, fatigue and balance disorders can be considered as the main concerns. Thus, gait restoration in patients with MS is the one of the primary objective of rehabilitation and often influences whether a patient can return home or to work. Even if potentially innovative treatments like treadmill training have been proposed, nowadays the role of robotic assisted locomotion rehabilitation has not been extensively studied in patients with MS.

DETAILED DESCRIPTION:
Background Multiple sclerosis (MS) is the most common chronic disabling disease of the central nervous system in young adults. Gait disorders represent one of the greatest causes of disability in patients with MS. Thus, gait restoration in patients with MS is the one of the primary objective of rehabilitation and often influences whether a patient can return home or to work.

Despite significant progress in the development of disease-modifying drugs, pharmacologic therapy alone does not warrant optimal care in MS. Exercise has been recognized as a feasible form of self-management for persons with the disease. Regular exercise can improve daily activity, cardiovascular fitness, muscle strength, health perception, and reduce fatigue in patients with MS.

To restore gait, modern concepts of rehabilitation support a repetitive task-specific approach. In recent years it has also been shown that higher intensities of walking practice (resulting in more repetitions trained) result in better outcomes for patients after stroke. Recently, the introduction of robotic devices for gait rehabilitation have showed to be a feasible approach in order to improve gait ability in patients with stroke and spinal cord lesions. These devices allow to train patients under a graduated body weight support condition and to guide the patient's steps reproducing a physiologic gait pattern for as long as the clinical conditions allow. This activity can be executed requiring only supervision by a physiotherapist and in absolutely safety condition for the patient.

Repetitive locomotor training is an innovative approach in gait disturbances in patients with multiple sclerosis. Only scant data on this issue is available and all these studies have been performed by means of conventional physiotherapy or treadmill training approaches. Nowadays the effectiveness of robotic devices for gait rehabilitation has not yet been evaluated in patients with multiple sclerosis.

Aim of the study The aim of the study is to evaluate the effect of a repetitive locomotor training by electromechanical gait trainer on gait endurance, fatigue and activities daily life in patients with MS.

Study Design Randomised controlled, blinded clinical trial. Materials and methods Fifty patients with definite diagnosis of MS according to McDonald criteria, and with EDSS score equal to or below 7 will be enrolled in the study. Patients with disease recurrence that worsens significantly during the 8 weeks before recruitment will be excluded. At the moment of recruitment (before treatment), at the end of treatment (6 weeks) and one month after the end of the treatment (FU) each patient will be tested with the following clinical and instrumental procedures. Clinical assessment procedures: 6-minute Walking Test, 10-meter Walking Test, Fatigue Severity Scale, Multiple Sclerosis Quality Of Life-54, Hamilton Rating Scale for Depression, Falls Efficacy Scale. Instrumental assessment procedures: GAITRite® System, Stabilometric Assessment and measure of energy cost by COSMED K4b2.

As primary outcome measure will be considered the 6-minute Walking Distance Test. As secondary outcomes measures will be considered the 10-meter Walking Test, Fatigue Severity Scale and the Multiple Sclerosis Quality Of Life-54, Hamilton Rating Scale for Depression, Falls Efficacy Scale, Spatio-temporal parameter with GAITRite® System, Stabilometric Assessment and measure of energy cost by COSMED K4b2. The allocation in the two groups will be done with simple randomisation.

Patients will be randomized into two groups. The first group (experimental group) will be subjected to 12 treatment session (2 sessions/week) on Gait Trainer machine. The second group (control group) will undergo to a conventional treatment with the same duration and frequency of the experimental group. Data will be analysed by means parametric and non-parametric tests. Both, within and between groups comparison will be performed. Data will be analyzed using SPSS software (ver 11.0; SPSS Inc., Chicago, IL, USA). Expected results: we could hypothesize that the training performed by the experimental group could improve gait endurance and daily life disability in patients with MS.

ELIGIBILITY:
Inclusion Criteria:

1. age between 30 and 60 years
2. Expanded Disability Status Scale (EDSS) score 2.0≥ x ≤ 4.0
3. Mini Mental State Evaluation (MMSE) score ≥ 24
4. absence of heart problems
5. ability to maintain standing position without aids for at least 1 minute
6. ability to walk independently for at least 15 metres
7. absence of concurrent neurological or orthopaedic diseases that interfere with deambulation.

Exclusion Criteria:

1. disease recurrence that worsens significantly during the 3 months prior to recruitment
2. pharmacological therapy not well defined
3. performance of any type of rehabilitation treatment in the month prior to recruitment
4. presence of other concurrent neurological or orthopaedic diseases involving the lower limbs and/or interfering with standing position and/or walking

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-11; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
6-minute Walking Test | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment and after the end (after 6 weeks) of the treatment.
  This is a validated test for the clinical evaluation of walking endurance using in patient with MS. It involves respiratory, cardiovascular, skeletal, nervous and muscular system competences/skills (32). The patient will be asked to walk at her/his self-selected walking speed in the gym along during the instrumental test.

SECONDARY OUTCOMES:
10-meter Walking Test | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
Falls efficacy scale score | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
  This is a scale used to assess fatigue in MS and other chronic diseases. It consists of a self-report questionnaire composed of nine items. Each item is scored on a seven-point scale ranging from 1 (absence of fatigue) to 7 (high level of fatigue). The score ranges from 9 to 63. Total score from each questionnaire will be reported in excel sheet at each evaluation session.
Spatio-temporal gait analysis | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
  Spatio-temporal gait analysis will be evaluated by using a computerized system called GAITRite system (Gold, version 3.2 b - CIR Systems, Inc, Havertown, PA). Patients will ask to ambulate along the 7.66m electronic walkway at their fastest speed. The following gait parameters will be considered: gait speed (cm/sec), cadence (step/min), stride length (cm), step length (cm), heel to heel base support (cm), swing of cycle (%), stance of cycle (%), single support of cycle (%) and double support of cycle (%). Each parameters will be reported in excel sheet at each evaluation session.
Static balance assessment | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
  The static balance assessment will be carried out with a monoaxial platform (Technoboby©) an electronic system used for the evaluation of the instant position of the centre of pressure (CoP), the length of CoP trajectory (LCop) and the distribution of sway area (DSA). The position of the feet on the platform is standardized using a V-shaped frame. The parameters above-mentioned will be calculated by computing data obtained under different visual conditions (eyes-open and eyes-closed) during a 30-sec time interval.
Measure of energy cost | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU
Hamilton Rating Scale for Depression | All patients enrolled in the study will be evaluated before the beginning (baseline time 0) of treatment, after the end (after 6 weeks) of the treatment and at 1 month FU

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Fiaschi, Professor, Study Chair — Department Neurological, Neuropsychological, Morphological and Movement Sciences, University of Verona, Verona, Italy
Locations (1):
- S.S.O. di Riabilitazione dell'Ospedale Policlinico, Verona, Verona, Italy

REFERENCES:
- [Background] Lo AC, Triche EW. Improving gait in multiple sclerosis using robot-assisted, body weight supported treadmill training. Neurorehabil Neural Repair. 2008 Nov-Dec;22(6):661-71. doi: 10.1177/1545968308318473. PMID 18971381
- [Background] Pohl M, Werner C, Holzgraefe M, Kroczek G, Mehrholz J, Wingendorf I, Hoolig G, Koch R, Hesse S. Repetitive locomotor training and physiotherapy improve walking and basic activities of daily living after stroke: a single-blind, randomized multicentre trial (DEutsche GAngtrainerStudie, DEGAS). Clin Rehabil. 2007 Jan;21(1):17-27. doi: 10.1177/0269215506071281. PMID 17213237
- [Background] Benedetti MG, Gasparroni V, Stecchi S, Zilioli R, Straudi S, Piperno R. Treadmill exercise in early mutiple sclerosis: a case series study. Eur J Phys Rehabil Med. 2009 Mar;45(1):53-9. PMID 19156023